CLINICAL TRIAL: NCT05069272
Title: A Randomized, Double-blinded, Vehicle Controlled, Monocentric Study to Evaluate the Efficacy and Tolerance of Synergistic Combination of Bakuchiol and Ethyl Linoleate on Mild to Moderate Acne Vulgaris
Brief Title: Double-blinded, Vehicle Controlled Study to Evaluate Efficacy & Tolerance of Bakuchiol and Ethyl Linoleate on Acne
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ratan K. Chaudhuri (Industry)
Responsible Party: Sponsor-Investigator, Ratan K. Chaudhuri, President, Sytheon Ltd.
Organization: Sytheon Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYTPIG1M
Record Dates: First submitted 2021-09-23; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — bakuchiol; ethyl linoleate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Synergistic combination of Bakuchiol and Ethyl Linoleate
  Interventions: Other: Bakuchiol and Ethyl Linoleate
- Vehicle (Placebo Comparator): No active ingredients
  Interventions: Other: Vehicle

INTERVENTIONS:
Other: Bakuchiol and Ethyl Linoleate — A synergistic combination of Bakuchiol and Ethyl Linoleate
  Arms: Intervention
Other: Vehicle — No actives
  Arms: Vehicle

SUMMARY:
Subjects will be assigned to a active cream or vehicle to compare the cosmetic effects. This will take place over a 12 week period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers, aged 18 years or older;
* with mild to moderate acne;
* Subjects must have between 10-100 non-inflammatory lesions and 10-50 inflammatory lesions but no more than 2 nodular lesions and no cysts on their face.
* If applicable, users of estrogens/birth control pills must have been on the treatment regimen for at least 3 months and be willing to continue use for study duration;

Females of child-bearing potential (FCBP): A female is considered not to be of childbearing potential if she is post-menopausal with at least 12 consecutive months of amenorrhea or has undergone surgical sterilization. While on the study, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

* Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR
* Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]; PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.
* Willing to follow study instructions and available to attend the study visits;
* Willing to provide written informed consent and sign photography release

Exclusion Criteria:

* Female subjects: Self-reported pregnant or breast feeding, or planning to become pregnant during the course of the study;
* Known allergy or hypersensitivity to acne treatment products;
* Current skin disease of any type in the test area (e.g. eczema, psoriasis, rosacea, seborrheic dermatitis, vitiligo, etc.), or under the treatment of a doctor for any skin condition;
* Have any cystic acne, acne conglobate, acne fulminans, or secondary acne (chloracne or drug-induced acne) in the test area;
* Any conditions on the test site that would interfere with evaluations (i.e. tattoos, scars, open cuts, sunburn, piercings, excessive hair, etc.);
* Use of topical treatments such as OTC (over the counter) acne medication topical anti-inflammatory medications, salicylic acid, corticosteroids, antibiotics, anti-bacterials, peroxide-containing products, or retinoids within 2 weeks of baseline;
* Use of depigmenting medications such as hydroquinone during the 14 days prior to the study start; Insulin dependent diabetes;
* Concurrent medication that might affect the response to the test articles including routine use of anti-inflammatory medications, anti-histamines, and steroids;
* History of Crohn's disease, or clinically significant enteritis (regional enteritis, ulcerative colitis, pseudomembranous colitis, antibiotic-associated colitis);
* Microdermabrasion or laser treatment in the test area within six months of the study;
* Medical condition which, in the opinion of the Investigator, would compromise the safety of the subject or confound study results;
* Use of systemic antibiotics, corticosteroids, antimalarials or oral dapsone within 4 weeks of baseline;
* Use of other anti-acne medications, including isotretinoin or spironolactone, within 6 months of baseline;
* Participation on an investigational drug study within 4 months of the baseline visit.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-02-20 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
IGA Score | From baseline to week 12
  IGA score of zero (clear) or one (almost clear)
Facial lesions | From baseline to week 12
  Percent reductions in facial lesion counts for inflammatory and noninflammatory

SECONDARY OUTCOMES:
Total lesion count | From baseline to week 2
  Percent change in Global Face Total Lesion Count
Total lesion count | From baseline to week 4
  Percent change in Global Face Total Lesion Count
Total lesion count | From baseline to week 8
  Percent change in Global Face Total Lesion Count
Total lesion count | From baseline to week 12
  Percent change in Global Face Total Lesion Count
IGA score | From baseline to week 2, 4, 8, 12
  IGA score of zero (clear) or one (almost clear) as compared to vehicle
IGA score | From baseline to week 4
  IGA score of zero (clear) or one (almost clear)
IGA score | From baseline to week 8
  IGA score of zero (clear) or one (almost clear)
IGA score | From baseline to week 12
  IGA score of zero (clear) or one (almost clear)
IGA score | From baseline to week 2, 4, 8 & 12
  IGA score of zero (clear) or one (almost clear) as compared to vehicle
Inflammatory and non-inflammatory leisons | From baseline to week 2
  Percent reductions in facial lesion counts for inflammatory and noninflammatory
Inflammatory and non-inflammatory leisons | From baseline to week 4
  Percent reductions in facial lesion counts for inflammatory and noninflammatory
Inflammatory and non-inflammatory leisons | From baseline to week 8
  Percent reductions in facial lesion counts for inflammatory and noninflammatory
Inflammatory and non-inflammatory leisons | From baseline to week 12
  Percent reductions in facial lesion counts for inflammatory and noninflammatory
Inflammatory and non-inflammatory leisons | From baseline to week 2, 4, 8 & 12
  Percent reductions in facial lesion counts for inflammatory and noninflammatory as compared to vehicle
Post inflammatory hyperpigmentation | From baseline to week 2
  Percent reduction in overall post inflammatory hyperpigmentation
Post inflammatory hyperpigmentation | From baseline to week 4
  Percent reduction in overall post inflammatory hyperpigmentation
Post inflammatory hyperpigmentation | From baseline to week 8
  Percent reduction in overall post inflammatory hyperpigmentation
Post inflammatory hyperpigmentation | From baseline to week 12
  Percent reduction in overall post inflammatory hyperpigmentation
Post inflammatory hyperpigmentation | From baseline to week 2, 4, 8 & 12
  Percent reduction in overall post inflammatory hyperpigmentation as compared to vehicle

CONTACTS AND LOCATIONS:
Overall Officials: Barrie Drewitt, Principal Investigator — Princeton Consumer Research
Locations (1):
- Princeton Consumer Research Corp, Chelmsford, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan on sharing IPD to other researchers